CLINICAL TRIAL: NCT00043212
Title: A Randomized, Double-blind, Placebo-controlled Phase III Clinical Trial Evaluating DCVax(tm)-Prostate, Autologous Dendritic Cells Loaded With Recombinant PSMA for the Treatment of Metastatic Hormone Refractory Prostate Cancer
Brief Title: Study of a Drug [DCVax (tm)-Prostate] to Treat Prostate Cancer When Hormone Therapy is no Longer Effective.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Redirection of company goals
Sponsor: Northwest Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DC3-HRPC, October 2001
Record Dates: First submitted 2002-08-06; First posted 2002-08-08 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; oncology; urology; hormone refractory prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

INTERVENTIONS:
Drug: Dendritic cell immunotherapy

SUMMARY:
The purpose of this clinical research study is to assess the safety and efficacy of an investigational therapy called DCVax(TM)-Prostate.

DETAILED DESCRIPTION:
Patients with hormone refractory prostate cancer are eligible if they have a rising PSA or three or fewer metastatic lesions. The experimental therapy uses a patient's own white blood cells and "teaches" the cells to recognize a "flag" on prostate cancer cells. This may help the immune system destroy prostate cancer cells. Side effects reported from the Phase I/II trial include skin reactions of redness, pain & swelling at the injection site, and short-lived headache, fever & fatigue. Full details are available in the informed consent.

ELIGIBILITY:
Inclusion Criteria

* Hormone refractory prostate cancer (HRPC) – progressive disease despite androgen deprivation and serum testosterone <50ng/dL; progression defined as either:

  1. Rising PSA over 6 months with at least a 50% increase between the 1st and 3rd measurement, and the 3rd measurement >2.0 ng/ml; or
  2. Progression of metastatic lesion on bone scan, or
  3. Progression of lymph node metastasis by CT scan.
* Zubrod or ECOG performance status of 0-1.
* Three or fewer bone metastases on a bone scan with minimal symptoms.
* No lymph node lesions greater than 3.0 cm at longest diameter.
* Adequate hematological, hepatic and renal function.

Exclusion Criteria

* History of other active malignancy.
* Prior chemotherapy, radiation therapy, immunosuppressive or investigational therapy for metastatic disease in previous 12 months.
* Strong opioids, immunosuppressives, megestrol acetate or other estrogenic hormones (e.g., Saw Palmetto, PC-SPES) within 1 month prior to enrollment.
* Brain, liver, or lung metastases; uncontrolled heart, liver, lung, or renal diseases or other serious illness.
* Prior splenectomy.
* History of severe asthma, anaphylaxis, or other serious adverse reactions to vaccines or any of the antigens included in the skin test.
* History of moderate to severe lower limb lymphedema, or recent signs of deep venous thrombosis (DVT) or thrombo-embolic disease, or impending stroke.
* History of immunodeficiency or autoimmune disease; positive HIV, HbsAg or anti-HCV.
* Impending untreated spinal cord compression or urinary outlet obstruction.
* Any medication that might affect immune function. (Exceptions: Nonprescription doses of NSAIDS; acetaminophen or aspirin; low doses of antihistamine therapy; normal range doses of vitamins; and H2 blockers).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Highlands Oncology Group, Springdale, Arkansas
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Diego Medical Center, San Diego, California
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Cancer Centers of Florida, P.A., Orlando, Florida
  - St. Francis Medical Center, Peoria, Illinois
  - Louisiana State University, New Orleans, Louisiana
  - Clinical Research Solutions, Las Vegas, Nevada
  - Albany Regional Cancer Center, Albany, New York
  - Carolinas HealthCare System, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Tyler Cancer Center, Tyler, Texas
  - University of Utah, Salt Lake City, Utah
  - Cancer Care Northwest, Spokane, Washington
  - St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- See also: Northwest Biotherapeutics, Inc. — http://www.nwbio.com